CLINICAL TRIAL: NCT00263419
Title: Psychosoziale Intervention Zur Reduktion Diabetischer Spätschäden Bei Diabetes Mellitus Typ 2
Brief Title: Stress-relief Management for Treatment of Late Complications in Type 2 Diabetes
Acronym: HEIDIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Stefan Kopf MD, Prof. P.P. Nawroth & Dr. med S. Kopf, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HD-Med1-01/05
Record Dates: First submitted 2005-12-07; First posted 2005-12-08 (Estimated); Last update posted 2011-10-27 (Estimated); Status verified 2011-10

CONDITIONS: Albuminuria; Diabetes Mellitus, Type 2; Diabetes Complications
Keywords: Diabetes Type 2; Late Complications; Stress relief management; psychosocial stress
MeSH Terms: conditions — Albuminuria; Diabetes Mellitus, Type 2; Diabetes Complications | interventions — Mindfulness-Based Stress Reduction

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction — 8 weeks mindfulness based stress reduction (MBSR) based on body and meditation practices that aims at cultivation of openness, awareness of the present moment and acceptance of all internal and external experiences. It is assumed that this allows to act more reflectively rather than impulsively.
  Other Names: Heidelberger Diabetes and Stress (HEIDIS) - Study

SUMMARY:
The purpose of this study is to determine whether a structured stress relief management program can prevent the progression of late diabetic complications in patients with type 2 diabetes.

DETAILED DESCRIPTION:
Patients with type 2 diabetes and increased albumin excretion have an increased risk of renal failure and cardiovascular events. It has recently been shown, that psychosocial stress is an additional major risk factor contributing to the increased risk of cardiac events. However, it is not clear, whether a structured stress-relief training of patients reduces the risk of micro- and macrovascular damage in type 2 diabetes.

Comparisons: Conventional treatment of diabetes according to national guidelines is compared to conventional treatment plus structured stress relief management training.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Type 2
* Albuminuria
* Age 30-70

Exclusion Criteria:

* Diabetes duration < 3 years
* Preexisting non-diabetic kidney
* Psychiatric disorders
* Alcohol or drug abuse
* Malignant tumors or hematologic disorders
* Heart failure NYHA III-IV
* Acute coronary syndrome

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2005-01; Primary Completion 2012-03 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Progression of albuminuria | 1,2,3,4 and 5 year

SECONDARY OUTCOMES:
Mortality | 3,4 and 5 years
Late diabetic complications (micro-macrovascular) | 1,2,3,4 and 5 years
Cardiovascular Events | 1, 2,3,4 and 5 years
Nuclear Factor kappa B as marker of psychosocial stress | 1,2,3,4 and 5 years
Quality of life | post intervention, 1,2,3,4 and 5 years
Psychological symptoms | post intervention, 1,2,3,4 and 5 years
Cardiovascular risk factors | post intervention, 1,2,3,4 and 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter P Nawroth, MD, Principal Investigator — University of Heidelberg, Dept. Medicine 1, Germany
Locations (1):
- Department of Medicine, University of Heidelberg, Heidelberg, Germany

REFERENCES:
- [Derived] Cashmore BA, Cooper TE, Evangelidis NM, Green SC, Lopez-Vargas P, Tunnicliffe DJ. Education programmes for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 Aug 22;8(8):CD007374. doi: 10.1002/14651858.CD007374.pub3. PMID 39171639
- [Derived] Kopf S, Oikonomou D, Hartmann M, Feier F, Faude-Lang V, Morcos M, Haring HU, Herzog W, Bierhaus A, Humpert PM, Nawroth PP. Effects of stress reduction on cardiovascular risk factors in type 2 diabetes patients with early kidney disease - results of a randomized controlled trial (HEIDIS). Exp Clin Endocrinol Diabetes. 2014 Jun;122(6):341-9. doi: 10.1055/s-0034-1372583. Epub 2014 May 5. PMID 24798861
- [Derived] Kopf S, Oikonomou D, von Eynatten M, Kieser M, Zdunek D, Hess G, Morcos M, Forsblom C, Bierhaus A, Groop PH, Nawroth PP, Humpert PM. Urinary excretion of high molecular weight adiponectin is an independent predictor of decline of renal function in type 2 diabetes. Acta Diabetol. 2014;51(3):479-89. doi: 10.1007/s00592-013-0542-2. Epub 2013 Dec 24. PMID 24366425
- [Derived] Hartmann M, Kopf S, Kircher C, Faude-Lang V, Djuric Z, Augstein F, Friederich HC, Kieser M, Bierhaus A, Humpert PM, Herzog W, Nawroth PP. Sustained effects of a mindfulness-based stress-reduction intervention in type 2 diabetic patients: design and first results of a randomized controlled trial (the Heidelberger Diabetes and Stress-study). Diabetes Care. 2012 May;35(5):945-7. doi: 10.2337/dc11-1343. Epub 2012 Feb 14. PMID 22338101